CLINICAL TRIAL: NCT06114563
Title: Effects of Yogurt With Spirulina Consumption in High Cardiometabolic Risk Individuals
Brief Title: Effects of Yogurt With Spirulina on Cardiometabolic Risk Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Collaborators: Hellenic Agricultural Organization DEMETER (Unknown)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Assistant Professor, Agricultural University of Athens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HRBD 41/26.05.2023
Record Dates: First submitted 2023-10-18; First posted 2023-11-02 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Overweight and Obesity; PreDiabetes; Hypertension; Dyslipidemias
Keywords: spirulina; yogurt; cardiometabolic risk factors
MeSH Terms: conditions — Overweight; Obesity; Prediabetic State; Hypertension; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spirulina yogurt (Experimental): 2 yogurts with spirulina each containing 2 g of spirulina
  Interventions: Other: Spirulina yogurt
- Conventional yogurt (Active Comparator): 2 conventional yogurts (without spirulina)
  Interventions: Other: Conventional yogurt

INTERVENTIONS:
Other: Spirulina yogurt — High cardiometabolic risk volunteers will be asked to consume 2 yogurts with spirulina, each containing 2 g spirulina, daily for 8 weeks, without any other change in their dietary habits and physical activity.
  Arms: Spirulina yogurt
Other: Conventional yogurt — High cardiometabolic risk volunteers will be asked to consume 2 conventional yogurts (without spirulina), daily for 8 weeks, without any other change in their dietary habits and physical activity.
  Arms: Conventional yogurt

SUMMARY:
The effects of yogurt with spirulina consumption compared to conventional yogurt (without spirulina) on several cardiometabolic and anthropometric parameters in individuals at risk of cardiovascular disease

DETAILED DESCRIPTION:
This randomized, double-blind, controlled clinical trial aims to evaluate the effects of the consumption of yogurt with spirulina compared to conventional yogurt in high cardiometabolic risk volunteers. Volunteers must be overweight/obese either with prediabetes, and/or hypertension, and/or hyperlipidemia and following a Westernized-type diet. The participants will be divided and randomly assigned into 2 groups. Each participant will be instructed to consume two 200 g servings of their designated low-fat sheep yogurt daily before consuming the main meal. The intervention group will receive two spirulina-enriched yogurt desserts daily, which will provide a total of 4 g spirulina per day, while the control group will receive unfortified yogurt along with their usual Westernized-type diet. Participants in both groups will be instructed to consume the two yogurts (enriched or plain), either all at once or separately, before their main meals, along with their usual Westernized diet. No other dietary advice will be provided to participants.

Participants will be asked to maintain their usual physical activity during the intervention period. At the beginning of the study, at 8 weeks, and 12 weeks after the beginning of the intervention (follow-up), blood samples will be collected after 12 hours of fasting. Two-hour oral glucose tolerance test (OGTT) will be performed using a continuous glucose monitoring system at the beginning and at 8 weeks. Blood lipids (total cholesterol, HDL-cholesterol, triglycerides, and LDL-cholesterol), CRP, IL-6, vitamin D, iron, ferritin, and total blood count will be measured at the beginning, 8 weeks, and 12 weeks. Anthropometric measurements (body weight and body composition analysis) will be performed at the beginning and every two weeks for 12 weeks. Basal metabolic rate (BMR) and central aortic blood pressure will be measured at the beginning, 4 weeks, 8 weeks, and 12 weeks of the intervention. Fecal samples will be collected and analyzed to study the gut microbiome composition at the intervention's beginning and at 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index >= 25 kg/m2
* Prediabetes [Fasting blood glucose > 100 mg/dL], or/and
* Hypertension [Systolic blood pressure (SBP) > 130 mmHg or Diastolic blood pressure (DBP) > 80 mmHg], or/and
* Hyperlipidemia [Total cholesterol > 200 mg/dL, and/or LDL-C > 100 mg/dL, and/or triglycerides > 150 mg/dL]

Exclusion Criteria:

* Severe chronic disease (e.g. cardiovascular diseases, diabetes mellitus, kidney or liver diseases, endocrine conditions)
* Medication that affects glycemia such as metformin, glucocorticoids, thiazide diuretics
* Gastrointestinal disorders
* Pregnancy
* Lactation
* Alcohol abuse
* Drug dependency
* Body weight lowering medications and/or history of bariatric surgery
* Depression and other psychiatric diseases
* Cancer
* Current spirulina intake

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Change in Fasting Blood Glucose Levels | Baseline, 8 weeks and 12 weeks outcome measurement (3 months)
  Blood glucose levels were determined at baseline, end of study, and at 12 weeks
Change in Total Cholesterol Levels | Baseline, 8 weeks and 12 weeks outcome measurement (3 months)
  Total cholesterol levels were determined at baseline, end of study, and at 12 weeks after dietary intervention
Change in HDL-cholesterol Levels | Baseline, 8 weeks and 12 weeks outcome measurement (3 months)
  HDL-cholesterol levels were determined at baseline, end of study, and at 12 weeks after dietary intervention
Change in LDL-cholesterol Levels | Baseline and end of 8 weeks and at 12 weeks follow-up outcome measurement (3 months)
  LDL-cholesterol levels were determined before diet intervention, at 8 weeks, LDL-cholesterol levels were determined at baseline, end of study, and at 12 weeks after dietary intervention
Systolic Blood Pressure | Baseline and end of 8 weeks and at 12 weeks follow-up outcome measurement (3 months)
  Systolic blood pressure levels were determined at baseline, end of study, and at 12 weeks after dietary intervention
Change in Triglyceride Levels | Baseline and end of 8 weeks and at 12 weeks outcome measurement (3 months)
  Triglyceride levels were determined before diet intervention, at 8 weeks, levels were determined at baseline, end of study, and at 12 weeks after dietary intervention
Diastolic Blood Pressure | Baseline and end of 8 weeks and at 12 weeks outcome measurement (3 months)
  Diastolic blood pressure levels were determined at baseline, end of study, and at 12 weeks after dietary intervention

SECONDARY OUTCOMES:
Change in energy intake | Baseline to 12 weeks (3 months)
  Change in energy intake (kcal/day) over the course of the study
Change in Blood Insulin Levels | Baseline and end of 8 weeks and at 12 weeks outcome measurement (3 months)
  Blood insulin levels were determined before diet intervention, at 8 weeks, and at 12 weeks after diet intervention
Oral Glucose Tolerance Test (OGGT) for Insulin Resistance Determination (Outcome Measures of Plasma Glucose Concentrations) | Outcome OGGT measurements performed before dietary intervention and after 8-week dietary intervention (2 months)
  Pharmacokinetic outcome measures: Determination of insulin resistance with OGGT testing. Before and after oral consumption of 75 g of glucose, capillary glucose concentrations were measured at the following times: 0 min - before oral consumption of 75 g glucose, 30 min, 60 min, 90 min, and 120 min after oral consumption of 75 g glucose
Change in basal metabolic rate (BMR) | Baseline to 12 weeks (3 months)
  Change in basal metabolic rate (kcal/day) over the course of the study
Change in central aortic blood pressure | Baseline to 8 weeks and to 12 weeks (3 months)
  Significant change in central pressure (mmHg)
Change in body weight | Baseline to 12 weeks (3 months)
  Change in body weight over the course of the study
Change in gut microbiome | Baseline to 8 weeks (2 months)
  The microbial composition in fecal samples will be measured via taxonomic profiling by 16S (V3-V4 region) ribosomal RNA gene amplicon sequencing using the MiSeq Illumina platform (v3 300bp pair-end sequencing) to identify a wide diversity of microbes
Time in target glucose range | Baseline to 8 weeks (2 months)
  Time spent in target glucose range of 70 to 180 mg/dL using FreeStyle Libre Continuous Glucose Monitor System
Glucose management indicator | Baseline to 8 weeks (2 months)
  Continuous glucose measurement (CGM) metric that indicates average blood glucose
Co-efficient of variation of glucose | Baseline to 8 weeks (2 months)
  CGM metric that measures variability in CGM values
Physical activity measures | Baseline to 12 weeks (3 months)
  Number of minutes of physical activity in the past week before visit
Change in Pulse Wave Velocity (PWV) | Baseline to 12 weeks (3 months)
  PWV using a noninvasive device was measured at baseline, 8 weeks, and 12 weeks after diet intervention
Change in C-reactive Protein levels | Baseline to 12 weeks (3 months)
  C-reactive Protein levels were measured at baseline, 8 weeks, and 12 weeks after diet intervention
Change in interleukin-6 (IL-6) levels | Baseline to 12 weeks (3 months)
  IL-6 levels were measured at baseline, 8 weeks, and 12 weeks after diet intervention
Change in vitamin D levels | Baseline to 12 weeks (3 months)
  vitamin D levels were measured at baseline, 8 weeks, and 12 weeks after diet intervention
Change in serum iron levels | Baseline to 12 weeks (3 months)
  Serum iron levels were measured at baseline, 8 weeks, and 12 weeks after diet intervention
Change in ferritin levels | Baseline to 12 weeks (3 months)
  Ferritin levels were measured at baseline, 8 weeks, and 12 weeks after diet intervention

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Papakonstantinou, PhD, Principal Investigator — Agricultural University of Athens
Locations (1):
- Agricultural University of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No